CLINICAL TRIAL: NCT05127083
Title: Oral Lichen Planus Photodynamic Treatment
Brief Title: Oral Lichen Planus Treatment
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universidad de Murcia (Other)
Responsible Party: Principal Investigator, Pia Lopez Jornet, Investigador principal Head Oral Medicine, Universidad de Murcia
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2227/2018
Record Dates: First submitted 2021-10-18; First posted 2021-11-19 (Actual); Last update posted 2021-11-19 (Actual); Status verified 2021-11

CONDITIONS: Oral Lichen Planus
Keywords: pain, oral lichen planus ; photodynamic therapy
MeSH Terms: conditions — Lichen Planus, Oral; Pain

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- toluidine blue-mediated photodynamic therapy (Experimental): The number of points will be variable according to the lesion size. Patients will be treated with localized PBM with a diode laser with continuous wave +toluidine blue
  Interventions: Radiation: Patients will be treated with localized PBM with a diode laser
- photodynamic therapy + gel (Active Comparator): The number of points will be variable according to the lesion size.atients will be treated with localized PBM with a diode laser with continuous wave
  Interventions: Radiation: Patients will be treated with localized PBM with a diode laser
- acetonide triamcinolone 0.2%+sham (Sham Comparator): Patients will be treated with acetonide triamcinolone 0.2% for 30 consecutive days. Laser device will be positioned over the lesion but will be switched off to mask the treatment. Patients will be instructed to apply the gel in the entire lesion three times/days.The number of points will be variable according to the lesion size.
  Interventions: Radiation: Patients will be treated with localized PBM with a diode laser

INTERVENTIONS:
Radiation: Patients will be treated with localized PBM with a diode laser — Toluidine blue was applied on the lesions.The tissue were irradiated with a 660-nm diode laser InGaAlP

SUMMARY:
Oral lichen planus (OLP) is a chronic inflammatory and immune-mediated disease affecting the oral mucosa. OLP presents with asymptomatic, lacelike white stripes and/or symptomatic red, ulcerated mucous membranes. Eating, drinking and oral hygiene procedures may be painful resulting in reduced quality of life (QOL). Photodynamic therapy (PDT) is a new suggestion for OLP treatment PDT is a successful treatment mo- dality for premalignant and malignant diseases of head and neck,gastrointestinal tract, lung, and skin

In this study, the effect of photodynamic therapy with topical corticosteroid in oral lichen planus patients was compared

DETAILED DESCRIPTION:
In this study, the efficacy of toluidine blue-mediated photodynamic therapy and topical triamcinolone acetonide 0.2% on decreasing pain and size of OLP lesions was compared.

This randomized, clinical trial compared the therapeutic effect of photodynamic therapy on symptomatic OLP (atrophic/ erosive/ulcerative forms) with triamcinolone acetonide 0.2%. The protocol of the clinical trial, which was conducted according to the ethical principles of Helsinki Group I toluidine blue-mediated photodynamic therapy Group II photodynamic therapy GroupIII laser sham + triamcinolone acetonide 0.2%

ELIGIBILITY:
Inclusion Criteria:

* . The patients with clinical or histopathological diagnosis of bilateral atrophic or erosive OLP (symptomatic OLP) who signed the written consent form were recruited.

Exclusion Criteria:

* Patients with drug-induced or contact lichenoid reactions, patients receiving any treatment for OLP in 2 months prior to the study, pregnant or lactating women, patients with uncontrolled systemic disease, and patients with photosensitivity

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2018-06-04 (Actual); Primary Completion 2020-10-03 (Actual); Study Completion 2021-10-18 (Actual)

PRIMARY OUTCOMES:
Change Assessment of Pain of OLP | Participants will be evaluated at baseline (Day 0) ; day 7: day 14 day and 28 day
  The pain will be assessed by applying a Visual Analog Scale, consisting of a 100-mm line numbered in centimeters, with two closed ends. One end is labeled "0" and the other "100", meaning no pain and terrible pain, respectively. Each patient will be instructed to mark a vertical line according to the best value that matches the intensity of pain during the evaluation.
Change Thongprasom sign scoring | Participants will be evaluated at baseline (Day 0) ; day 7: day 14 day and 28 day
  a score of 0 for normal healthy mucosa, 1 for lesions with only white striae, 2 for mixed keratotic and atrophic or erythematous lesions < 1 cm2 in size, 3 for keratotic and atrophic or erythematous lesions more than 1 cm2 in size, 4 for erosive/ulcerative lesions smaller than 1 cm2 , and 5 for erosive/ulcerative lesions larger than 1 cm2

CONTACTS AND LOCATIONS:
Locations (1):
- Lopez-Jornet Pia, Murcia, N/A = Not Applicable, Spain

IPD SHARING:
Plan to Share IPD: Yes

REFERENCES:
- [Background] Lavaee F, Shadmanpour M. Comparison of the effect of photodynamic therapy and topical corticosteroid on oral lichen planus lesions. Oral Dis. 2019 Nov;25(8):1954-1963. doi: 10.1111/odi.13188. Epub 2019 Oct 2. PMID 31478283
- [Background] Hoseinpour Jajarm H, Asadi R, Bardideh E, Shafaee H, Khazaei Y, Emadzadeh M. The effects of photodynamic and low-level laser therapy for treatment of oral lichen planus-A systematic review and meta-analysis. Photodiagnosis Photodyn Ther. 2018 Sep;23:254-260. doi: 10.1016/j.pdpdt.2018.07.001. Epub 2018 Jul 10. PMID 30006319
- [Background] Mostafa D, Moussa E, Alnouaem M. Evaluation of photodynamic therapy in treatment of oral erosive lichen planus in comparison with topically applied corticosteroids. Photodiagnosis Photodyn Ther. 2017 Sep;19:56-66. doi: 10.1016/j.pdpdt.2017.04.014. Epub 2017 Apr 25. PMID 28450262
- [Background] Rakesh N, Clint JB, Reddy SS, Nagi R, Chauhan P, Sharma S, Sharma P, Kaur A, Shetty B, Ashwini S, Pavan Kumar T, Vidya GS. Clinical evaluation of photodynamic therapy for the treatment of refractory oral Lichen planus - A case series. Photodiagnosis Photodyn Ther. 2018 Dec;24:280-285. doi: 10.1016/j.pdpdt.2018.09.011. Epub 2018 Sep 24. PMID 30261326
- [Derived] Salinas-Gilabert C, Gomez Garcia F, Galera Molero F, Pons-Fuster E, Vander Beken S, Lopez Jornet P. Photodynamic Therapy, Photobiomodulation and Acetonide Triamcinolone 0.1% in the Treatment of Oral Lichen Planus: A Randomized Clinical Trial. Pharmaceutics. 2022 Dec 22;15(1):30. doi: 10.3390/pharmaceutics15010030. PMID 36678659